CLINICAL TRIAL: NCT03368339
Title: Effectiveness of PR013 Topical Ophthalmic Drops Compared to Vehicle of PR013 Topical Ophthalmic Drops for the Treatment of Allergic Conjunctivitis Using Conjunctival Allergen Challenge Model (Ora-CAC®)
Brief Title: Effectiveness of PR013 Topical Ophthalmic Drops Compared to Vehicle for the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Realm Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-100-0007
Record Dates: First submitted 2017-11-20; First posted 2017-12-11 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-08

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PR013 topical Ophthalmic Drops (0.045%) (Active Comparator): topical Ophthalmic Drops (0.045%)
  Interventions: Drug: PR013 (0.045%)
- PR013 topical Ophthalmic Drops (0.06%) (Active Comparator): topical Ophthalmic Drops (0.06%)
  Interventions: Drug: PR013 (0.06%)
- Vehicle (Placebo Comparator): Placebo
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: PR013 (0.045%) — PR013 topical Ophthalmic Drops (0.045%)
  Other Names: HOCl
  Arms: PR013 topical Ophthalmic Drops (0.045%)
Drug: PR013 (0.06%) — PR013 topical Ophthalmic Drops (0.06%)
  Other Names: HOCl
  Arms: PR013 topical Ophthalmic Drops (0.06%)
Drug: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
To evaluate the efficacy and safety of PR013 topical ophthalmic drops (0.045% and 0.06%) compared to vehicle for the treatment of the signs and symptoms of allergic conjunctivitis using a modified Conjunctival Allergen Challenge Model (Ora-CAC®).

DETAILED DESCRIPTION:
A Multi-Center, Double-Masked, Randomized, Phase 2 Evaluation of the Effectiveness of PR013 Topical Ophthalmic Drops (0.045% and 0.06%) Compared to Vehicle of PR013 Topical Ophthalmic Drops for the Treatment of Allergic Conjunctivitis Using a Modified Conjunctival Allergen Challenge Model (Ora-CAC®)

ELIGIBILITY:
Inclusion Criteria:

* be at least 10 years of age of either sex and any race
* have a positive history of ocular allergies and a positive skin test reaction to a perennial allergen (cat dander, dog dander, dust mites, cockroaches) and a seasonal allergen (trees, grasses, and/or ragweed) as confirmed by an allergic skin test within the past 24 months.
* have a calculated visual acuity of 0.7 logMAR or better in each eye as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart

Exclusion Criteria:

* have known contraindications or sensitivities to the use of the investigational product or any of its components
* have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium or a diagnosis of dry eye)
* have had ocular surgical intervention within 3 months prior to Visit 1 or during the study and/or a history of refractive surgery within the past 6 months
* have a known history of retinal detachment, diabetic retinopathy, or active retinal disease
* have the presence of an active ocular infection (bacterial, viral or fungal) or positive history of an ocular herpetic infection at any visit
* use any of the disallowed medications* during the period indicated prior to Visit 1 and during the study
* have any significant illness (e.g. any autoimmune disease requiring therapy, severe cardiovascular disease [including arrhythmias] the investigator feels could be expected to interfere with the subject's health or with the study parameters and/or put the subject at any unnecessary risk (includes but is not limited to: poorly controlled hypertension or poorly controlled diabetes, a history of status asthmaticus, organ transplants, a known history of persistent moderate or severe asthma, or a known history of moderate to severe allergic asthmatic reactions to any of the study allergens;
* have planned surgery (ocular or systemic) during the trial period or within 30 days after;
* have used an investigational drug or medical device within 30 days of the study or be concurrently enrolled in another investigational product trial;
* be a female who is currently pregnant, planning a pregnancy, or lactating

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
Ocular itching evaluated by the subject | [Time Frame: Efficacy assessment period (Day 7 through Day 8)]
  The method of assessment for this outcome is the Ora Calibra(TM) Conjunctival Allergen Challenge Ocular Itching Scale
Conjunctival redness evaluated by the Investigator | [Time Frame: Efficacy assessment period (Day 7 through Day 8)]
  Ora Calibra(TM) Ocular Hyperemia Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Cesano, MD, Study Chair — Essa Pharma
Locations (1):
- Principal Investigator, Philadelphia, Pennsylvania, United States